CLINICAL TRIAL: NCT01805245
Title: Mindfulness: a Novel Approach for the Management of Diabetes-related Distress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 11-0333
Record Dates: First submitted 2012-06-15; First posted 2013-03-06 (Estimated); Last update posted 2017-04-19 (Actual); Status verified 2017-04

CONDITIONS: Emotional Distress; Type 2 Diabetes; Stress
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mindfulness Based Stress Reduction (Experimental)
  Interventions: Behavioral: Mindfulness Based Stress Reduction
- Health Education Control (Active Comparator)
  Interventions: Behavioral: Mindfulness Based Stress Reduction

INTERVENTIONS:
Behavioral: Mindfulness Based Stress Reduction — Standard 8-week MBSR program; classes meet for 2.5 hours once weekly The health education control group meets at the same time and for the same amount of time

SUMMARY:
The purpose of this study is to evaluate the impact of stress reduction on physiological and psychological variables in adults with Type 2 diabetes (T2DM) who have moderate to severe levels of diabetes-related emotional distress. Subjects will be randomized to one of two interventions. We will evaluate the impact of the interventions on glucose metabolism, blood pressure, diabetes-related distress and quality of life. Additionally, we will investigate the role of neuroendocrine dysfunction, systemic inflammation and diabetes self-care practices as mediators in the relationship between increased stress, adverse glucose metabolism and elevated blood pressure in those subjects with T2DM.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 30 years
2. Male or female
3. Duration of diabetes 1-15 years from time of initial diagnosis
4. Diagnosis of T2DM made/confirmed by physician
5. Completed diabetes education in the past
6. Most recent HgA1c >7%; measurement must be within the past 6 months either in physicians office or at the Thriving with Diabetes Boot Camp Class
7. Treatment for diabetes must include any or all of the following modalities:

   diet, exercise, oral medications, insulin or other injectable diabetic medication
8. Score > 30 on the Problem Area in Diabetes (PAID) Questionnaire
9. Able to use a glucometer for self-monitoring of blood glucose values
10. Most recent clinic blood pressure less than 180/95

Exclusion Criteria:

1. History of ketoacidosis
2. Age at diagnosis of T2DM < 30 years
3. Score >15 on the PHQ-9
4. Previous training in relaxation or meditation techniques
5. Current practice of yoga, tai chi or any other mind-body movement for > 60 minutes per week
6. Current use of a psychoactive drug for less than 3 months or not yet on a stable dose
7. Inability to participate fully or behave appropriately in the group treatment setting, as observed by baseline acknowledgement of substance abuse, psychotic episode(s), psychiatric hospitalization or history of self- harm within the past 2 years, or current suicidal or homicidal ideation
8. Inability to complete standardized instruments because of a cognitive deficit or language barrier
9. Current use or use within the past 3 months of oral glucocorticoids, excluding intraocular, topical or inhaled preparations
10. History of inflammatory diseases including rheumatoid arthritis and inflammatory bowel disease
11. Use of immune modulating agents
12. Night shift work or other type of schedule in which sleep wake cycle is disrupted
13. Women who consume > 7 alcoholic drinks per week and men who consume > 14 drinks per week
14. Current use or history of daily tobacco use within the past 1 year
15. End stage renal failure on dialysis
16. Pregnancy or post partum <3 months
17. Subjects with known secondary causes of hypertension including renal artery stenosis, pheochromocytoma, coarctation of aorta, hyperaldosteronemia
18. Non-dominant arm circumference > 46cm
19. Unwilling to accept randomization

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2012-01; Primary Completion 2014-11 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
HgA1c | 0,8,24 weeks
  We will assess change in glycemic control using the A1c. It will be measured at baseline, immediately following the 8 week intervention and at 24 weeks from baseline.
Diabetes Distress | 0,8,24 weeks
  The Problem Areas in Diabetes will be used to assess the change in diabetes emotional distress at baseline, immediately following the 8 week intervention and at 24 weeks from baseline

SECONDARY OUTCOMES:
SF36 Physical Health Score | 0, 8,24 weeks
  This measure is a patient reported outcome assessing general quality of life and will be assessed using the standardized SF36 tool.
SF36 Mental Health Score | 0,8,24 weeks
  This measure is a patient reported outcome assessing general quality of life and will be assessed using the standardized SF36 tool.
Mean 24 hour ambulatory systolic blood pressure | 0,8,24 weeks
  Mean systolic blood pressure over 24 hours.
Mean 24 hour diastolic ambulatory blood pressure | 0,8,24 weeks
  Mean diastolic blood pressure over 24 hours
HOMA-IR | 0,8,24 weeks
  For those participants that are not using insulin, we will assess the degree of insulin resistance using the HOMA-IR, which is derived from the fasting insulin and fasting glucose.
Depression | 0,8,24 weeks
  Using the Beck Depression Inventory we will assess symptoms of depression using this standardized patient reported outcome.
State Anxiety | 0,8,24 weeks
  Using the State and Trait Anxiety Assessment we will measure "state" anxiety.
Trait Anxiety | 0,8,24 weeks
  Using the State and Trait Anxiety Survey we will assess "trait" anxiety.
Social Support | 0,8,24 weeks
  Using the Duke Social Support and Stress Scale we will assess the degree of social support participants report in their lives.
Coping Style | 0,8,24 weeks
  Using the Coping Orientation to Problems Experienced Scale, we will evaluate the various coping styles and how they may change over time.
General Stress | 0,8,24 weeks
  Using the Perceived Stress Scale we will assess general life stressors.
Cortisol 24 hour area under the curve | 0,8,24 weeks
  Calculating the area under the curve for 24 hours we will assess cortisol secretion as a physiological assessment of stress
Cortisol Awakening Response | 0,8,24 weeks
  We will measure the cortisol awakening response using measures of cortisol prior to arising and 30 minutes after waking up.
IL-6 | 0,8, 24 weeks
  IL-6 is an assessment of systemic inflammation and will be measured in serum.
Summary of Diabetes Self-Care Activities | 0,8,24 weeks
  This patient reported measure assesses the frequency which participants engage in self-care activities that are critical for DM self-management.
Average 24 hour glucose by continuous glucose monitor (cgm) | 0,8,24 weeks
  Average cgm glucose over 24 hours
Average night time glucose | 0,8,24 weeks
  Average night time glucose from 10pm-6am using continuous glucose monitoring values
Average day time glucose | 0,8,24 weeks
  Average day time glucose from 6am-10pm using continuous glucose monitoring values
Block Food Frequency Questionnaire | Week 0
  Standardized assessment of dietary patterns
Mean Day Systolic Ambulatory Blood Pressure | 0,8,24 weeks
  The average systolic blood pressure measured by ambulatory blood pressure monitoring between 6 am and 10 pm
Mean Day Diastolic Ambulatory Blood Pressure | 0,8,24 weeks
  The average systolic blood pressure measured by ambulatory blood pressure monitoring between 6 am and 10 pm
Mean Night Systolic Ambulatory Blood Pressure | 0,8,24 weeks
  The average systolic blood pressure measured by ambulatory blood pressure monitoring between 10 pm and 6 am.
Mean Night Diastolic Ambulatory Blood Pressure | 0,8,24 weeks
  The average diastolic blood pressure measured by ambulatory blood pressure monitoring between 10 pm and 6 am.

OTHER OUTCOMES:
Mindfulness | 0,8,24 weeks
  To assess mindfulness we will utilize the Five Facet Mindfulness Questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Laura A Young, MD, PhD, Principal Investigator — University of North Carolina
Locations (1):
- University of North Carolina, Chapel Hill, North Carolina, United States